CLINICAL TRIAL: NCT07386184
Title: Histological and Radiological Evaluation of Collagenic Porcine Graft vs Collagen-enriched Bovine-derived Graft in Transcrestal Sinus Elevation. A Randomized Prospective, Controlled Study.
Brief Title: Collagenic vs Collagen-enriched Graft in Sinus Elevation: RCT
Acronym: C vs CE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Responsible Party: Principal Investigator, Luigi Canullo, professor, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SINUS 2
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sinus Lift Augmentation
Keywords: Randomized controlled prospective clinical trial

STUDY DESIGN:
Intervention Model Description: All patients will undergo the same intervention (sinus lift with crystal approach) using two different graft materials
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- insertion of porcine collagenic graft in the sinus (Experimental): porcine graft, which, due to its deantigenation process, results to be completely enbibed with its native collagen. This was demonstrated to allow a better regeneration due to its angiogenic and osteogenic potential
  Interventions: Procedure: transcrestal sinus lift
- bovine collagen enriched graft (Active Comparator): the collagen-enriched bovine-derived bone substitute is composed predominantly of deproteinized bovine bone granules combined with a minor fraction of highly purified porcine collagen. The addition of collagen improves the handling properties and moldability of the graft, facilitating its clinical application.
  Interventions: Procedure: transcrestal sinus lift

INTERVENTIONS:
Procedure: transcrestal sinus lift — Transcrestal sinus floor elevation (tSFE) is a surgical technique released through the use of guided surgery and specifically designed drills aimed to release the sinus mucosa. The use of micro elevators is aimed to detach the mucosa from the bone and free the space for the graft material. Graft material is inserted using specific pluggers.

SUMMARY:
The goal of this clinical trial is to histologically understand if collagenic or collagen enriched graft in sinus lift of healthy volunteers needing for implants in the posterior maxillae may work. The main question it aims to answer are:

which material works better histologically and radiologically? Researchers will compare a collagenic graft to collagen enriched graft to see if the osteointegration of the material is the same.

Participants will undergo a sinus lift with one of the two materials and after six month will undergo a bone sample collection to allow the implant insertion.

twelve moths thereafter, a radiograph will be taken to measure the extension of the bone regeneration and implant behavior

DETAILED DESCRIPTION:
Transcrestal sinus floor elevation (tSFE) is an established technique for vertically augmenting bone in the edentulous posterior maxilla, offering a less invasive alternative to the lateral approach.

Among the various bone substitutes used in transcrestal sinus augmentation, one widely adopted option is the collagen-enriched bovine-derived bone substitute. This material is composed predominantly of deproteinized bovine bone granules combined with a minor fraction of highly purified porcine collagen. The addition of collagen improves the handling properties and moldability of the graft, facilitating its clinical application.

An alternative approach involves the use of porcine graft, which, due to its deantigenation process, results to be completely enbibed with its native collagen. This was demonstrated to allow a better regeneration due to its angiogenic and osteogenic potential The primary objective of the present study is to perform a histological evaluation of the quality of bone regeneration following the placement of a graft material during transcrestal sinus floor elevation in cases of severely resorbed posterior maxilla. Specifically, the analysis will quantify the relative proportions of native bone, newly formed bone, connective tissue, and residual graft material within the augmented area. The secondary objectives are to assess, through radiographic analysis, the volumetric changes of the grafted area over time-including the rate of graft material resorption or shrinkage-and to evaluate the implant survival rate associated with this regenerative approach.

Materials and Methods: The study was designed as a prospective, randomized, controlled clinical trial. All patients requiring an implant-supported restoration in the posterior maxilla with a residual bone height of less than 4 mm beneath the maxillary sinus floor were eligible for the study. A minimum sample of 12.2 participants for each group (24.4 participants in total) was required to detect significant differences between the two groups Preoperatively, all patients will undergo a comprehensive clinical and radiographic evaluation. This includes a full periodontal examination, assessment of occlusal relationships, and evaluation of the prosthetic space. Cone Beam Computed Tomography (CBCT) scans and digital dental impressions will be obtained. The resulting Standard Tessellation Language (STL) and Digital Imaging and Communications in Medicine (DICOM) files will be matched and integrated into a digital workflow for virtual planning using dedicated software (RealGUIDE, 3DIEMME, Cantù, Italy).

Following the administration of local anesthesia (2% mepivacaine HCl with 1:100,000 epinephrine), a minimally invasive full-thickness envelope flap will be elevated to expose the surgical site. Access to the sinus cavity will be achieved via a crestal approach. Initial drilling will be performed using a 2 mm drill until contact with the cortical bone of the sinus floor. Subsequently, osteotomic screws of increasing diameters (typically 3.5 and 4.0 mm) will be used to complete the crestal antrostomy. A preliminary detachment of the Schneiderian membrane will be performed using specially designed microelevators (Dajelevators, Merighi Umberto, Valsamoggia, Italy). After checking membrane integrity using the Valsalva maneuver, the selected bone graft material will be inserted in small increments and gently compacted using a plugger to further elevate the sinus membrane from the floor and the lateral and medial walls of the sinus cavity. Collagenic porcine bone graft (MP3, Osteobiol, Giaveno, Italy) will be inserted in test group, while a collagen-enriched, bovine-derived bone substitute (Bio-Oss Collagen, Geistlich, Wolhusen, Switzerland) will be used in the control group. Once a satisfactory elevation will be achieved-defined as a total height of at least 10 mm from the crestal bone level to the elevated membrane position, as verified by intraoperative periapical radiographs-the crestal access will be sealed with a final increment of graft material.

The flap will be then closed using resorbable 6-0 sutures (Monofast, Medipac, Greece), using single interrupted stitches. Postoperative care included a 5-day antibiotic regimen (amoxicillin/clavulanate 1 g three times daily) and nonsteroidal anti-inflammatory medication (ketoprofen 80 mg as needed). Sutures will be removed after 14 days, and healing will be monitored on a monthly basis.

A CBCT scan will be performed to assess the tridimensional integrity of the mucosal elevation.

Dental implants installation and prosthetics. After a 6-month healing period, a CBCT scan will be performed to assess the quality and maturation of the regenerated tissue. Subsequently, dental implants will be placed according to the pre-established surgical plan. Following local anesthesia and minimally invasive flap elevation, a surgical stent will be used to guide the osteotomy. A 4 mm external diameter trephine bur, mounted on a surgical motor (SA-310 Elcomed, W&H, Bürmoos, Austria) will be used to harvest a bone core from the planned implant site. The retrieved bone specimens will be immediately immersed in 10% buffered formalin solution (Carlo Erba Reagents, Cornaredo, Italy) for histological analysis. The implant osteotomy will be then completed, and the implants were inserted as planned.

After an additional 4-month healing period, prosthetic rehabilitation will be performed following standard clinical protocols.To assess dimensional changes in the grafted area, preoperative, immediately post operative and 6-month postoperative CBCT scans will be analyzed. Variations in the augmented region will be evaluated in terms of bone height and graft volume. For linear measurements, the implant site will be used as a reference, and assessments will be performed along the ideal implant axis, previously determined using 3D planning software. Crestal bone height (CBH) will. be defined as the vertical distance between the alveolar crest and the sinus floor.

Sinus width will be measured as the medio-buccal dimension at 10 mm from the crest. A threshold of 12 mm will be used to define the sinus as either wide (>12 mm) or narrow (≤12 mm). For volumetric analysis, three-dimensional reconstructions of the grafted areas will be obtained using a semi-automatic segmentation protocol performed in 3D Slicer (version 5.2.1), an open-source software platform for medical image analysis.Segmentation will be carried out by an experienced operator using a combination of threshold-based and manual refinement techniques. For each implant site, a STL file of the grafted volume will be generated. STL files will be then processed using MeshLab (version 2023.12), an open-source system for 3D mesh processing (www.meshlab.net) to calculate the total graft volume, expressed in cubic millimeters (mm³).Bone samples will be fixed in 10% buffered formalin (Carlo Erba Reagents, Cornaredo, Italy) immediately after harvesting to minimize tissue alterations. Fixation will be carried out for 72 hours, followed by a thorough rinse in water to remove residual formalin. Samples will be then decalcified in 17% EDTA, pH 10 (Carlo Erba Reagents, Cornaredo, Italy) using a microwave-assisted protocol, as previously described (Savadori et al., 2023). The endpoint of decalcification will be determined using the ammonium oxalate chemical test (Giardino et al., 2019). After decalcification, specimens will undergo dehydration in a graded ethanol series (70% to 100%), xylene clarification, and paraffin embedding (Giardino et al., 2023). Histological sections 4 μm thick will be obtained using a rotary microtome (RM2245, Leica Biosystems, Nussloch, Germany). Only sections derived from the central portion of each biopsy, thereby avoiding areas potentially affected by friction from the trephine bur, will be included in the analysis. Sections will be mounted on silanized glass slides (VWR International, Radnor, PA, USA) and stained with hematoxylin and eosin (Carlo Erba Reagents, Cornaredo, Italy) to enable identification and quantification of newly formed bone and residual biomaterial, as well as qualitative assessment of soft tissue morphology, cellular composition, and inflammatory response.

Images will be acquired using a transmitted light microscope (CX43, Olympus Corporation, Tokyo, Japan) equipped with an Olympus LC30 camera and processed with LCmicro software (version 2.2) (Olympus Corporation, Tokyo, Japan). For each sample, three representative sections will be analyzed. Multiple high-resolution micrographs will be taken per section and digitally stitched into a single panoramic image using AutoStitch software (version 1.0) (University of British Columbia, Vancouver, Canada; www.cs.ubc.ca/~mbrown/autostitch/autostitch.html). These composite images will be used for histomorphometric analysis to quantify the areas of newly formed bone and residual biomaterial, expressed as a percentage of the total section area. Measurements will be performed on all three sections, and the arithmetic mean was calculated. Image analysis will be carried out using ImageJ software (National Institutes of Health, Bethesda, MD, USA; https://imagej.nih.gov/ij/). The same images will be also used for qualitative evaluation.

For standardized analysis, each bone core will be divided into 2.5 mm-long segments, to avoid comparing areas with different regenerative patterns within the same plane, and to reduce potential bias caused by core fractures during harvesting or processing. Although efforts will be made to obtain cores of uniform length (7-8 mm), there is the possibility that intact samples will be not always retrievable due to mechanical fragility during trephine extraction or decalcification. For this reason, the segmental analysis approach will be adopted as the methodological standard: poorly mineralized samples, in which only a limited segment could be evaluated, will be thus not weighted equally to longer, structurally intact specimens. Non-regenerated portions will be excluded from analysis when their mechanical integrity is compromised.

In addition, hematoxylin and eosin (H&E) staining will be used for a semi-quantitative assessment of inflammatory infiltrates, based on a previously validated scoring system. Inflammatory response will be graded according to the density and distribution of inflammatory cells, as follows:

* Score 0: No inflammatory infiltrate
* Score 1: Occasional isolated mononuclear cells
* Score 2: Focal mononuclear infiltrate with limited distribution
* Score 3: Diffuse mononuclear infiltrate of moderate intensity
* Score 4: Extensive infiltrate with cellular aggregates and/or granulocytic components.

Statistical analysis and data visualization will be performed using GraphPad Prism (version 8.0.1 for Windows; GraphPad Software, Boston, MA, USA). All variables in the dataset will be first tested for normality using the Shapiro-Wilk test. Data will be then summarized using mean and standard deviation for normally distributed variables, or median and interquartile range (IQR) for non-normally distributed variables.

Differences between the test and control groups in terms of age, residual crestal bone height, sinus medio-buccal dimension, total mineralized tissue, newly formed bone, residual graft, and mesh volume (mm³) will be assessed using either the unpaired t-test or the Mann-Whitney U test, depending on the normality of distribution. Differences in categorical variables (gender, smoking habits, history of periodontitis, presence of membrane perforation) will be assessed using the Fisher's exact test. Intergroup differences in the mean ranks of newly formed bone and residual graft across the three defined regions of the bone core will be analyzed using the Kruskal-Wallis test.

For all statistical analyses, a p-value ≤ 0.05 was considered statistically significant. The null hypothesis in each case stated that there will be no difference between groups for the parameter being tested.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring vertical elevation of the maxillary sinus floor.
* Residual alveolar bone height of edentulous maxilla below the floor of the maxillary sinus <5 mm.
* Males and females between 30-80 years old
* Patients with healthy periodontal conditions (treated periodontitis, PI<25%, BoP<25%).
* Patients willing to sign an informed consent and participate in a clinical study.
* Generally fit and healthy and able to undergo oral surgical procedures under local anesthesia.
* Teeth at the surgical site requiring extraction were removed at least 12 weeks prior to sinus floor elevation.

Exclusion Criteria:

* Patients who smoke more than 5 cigarettes/day
* Pregnancy (confirmed by verbal inquiry)
* Chronic systemic pathologies (e.g. diabetes) and neoplasms of the oro-facial district.
* Patients undergoing treatment with antiresorptive agents.
* Patients receiving systemic corticosteroid therapy.
* Any site with a history of implant failure.
* Dental sites with acute infections.
* Chronic inflammatory diseases of the oral cavity.
* Autoimmune diseases.
* Documented hypersensitivity to any of the medications intended for use during the treatment protocol.
* Substance abusers.
* Patients with known collagen hypersensitivity.
* Patients with hypersensitivity to porcine-derived materials.
* History of malignant tumors of the maxillary sinus.
* History of head/neck radiation therapy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
histomorphometric analysis | 6 months
  For standardized analysis, each bone core will be divided into 2.5 mm-long segments. Although efforts will be made to obtain cores of uniform length (7-8 mm), there is the possibility that intact samples will be not always retrievable due to mechanical fragility during trephine extraction or decalcification. For this reason, the segmental analysis approach will be adopted as the methodological standard: poorly mineralized samples, in which only a limited segment could be evaluated, will be thus not weighted equally to longer, structurally intact specimens. Non-regenerated portions will be excluded from analysis when their mechanical integrity is compromised.
  Percentage of regenerated bone, native bone, graft, connective tissue will be measure
histologic analysis | 6 months
  Hematoxylin and eosin (H&E) staining will be used for a semi-quantitative assessment of inflammatory infiltrates, based on a previously validated scoring system.Additionally, immunohistochemistry (Osteolcin, Osteopontin, Osteonectin, RUNX2, TRAP, PAS) and Herovici, Sirius Red, RGB Trichrome will be run.

SECONDARY OUTCOMES:
linear radiologic measures | 12 months
  To assess dimensional changes in the grafted area, preoperative, immediately post operative and 6-month postoperative CBCT scans will be analyzed. Variations in the augmented region will be evaluated in terms of bone height and graft volume. For linear measurements, the implant site will be used as a reference, and assessments will be performed along the ideal implant axis, previously determined using 3D planning software. Crestal bone height (CBH) will. be defined as the vertical distance between the alveolar crest and the sinus floor.
  Sinus width will be measured as the medio-buccal dimension at 10 mm from the crest. A threshold of 12 mm will be used to define the sinus as either wide (>12 mm) or narrow (≤12 mm). Sinus width will be measured as the medio-buccal dimension at 10 mm from the crest. A threshold of 12 mm will be used to define the sinus as either wide (>12 mm) or narrow (≤12 mm).
3D radiologic measures | 12 months
  For each implant site, a STL file of the grafted volume will be generated. STL files will be then processedto calculate the total graft volume, expressed in cubic millimeters

IPD SHARING:
Plan to Share IPD: No
personal data sensibility.